CLINICAL TRIAL: NCT04716413
Title: Evaluating the Use of Sublingual Sufentanil in Patients With Suboxone Treatment Who Are Undergoing Ambulatory Surgery- a Case Series
Brief Title: Evaluating the Use of Sublingual Sufentanil in Patients With Suboxone Treatment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated early due to funding, lack of participants
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-12649
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Dsuvia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Subjects will receive dose of Dsuvia 30mcg SL (1st dose) after induction but before first incision. Post-operatively, if subject rates pain higher than 4 out of 10, subject will receive a second dose of Dsuvia 30mcg SL (sublingual). If 30 minutes after second dose, subject rates pain higher than 4 out of 10, subject will receive ibuprofen 800mg IV. If 60 minutes after second dose, subject rates pain higher than 7 out of 10, subject will receive hydromorphone 0.4 mg IV.
  Interventions: Drug: Dsuvia
- Control (No Intervention): Subjects will be receive routine standard of care.

INTERVENTIONS:
Drug: Dsuvia — Subject will receive up to 2 doses of Dsuvia. The first dose will be intra-op and the second dose will be post-op (if needed)
  Arms: Treatment

SUMMARY:
In this case series study, the investigators are testing the hypothesis that sublingual sufentanil (Dsuvia) will improve postoperative pain management in the Post Anesthesia Care Unit (PACU) in ambulatory surgery patients taking Suboxone.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-100 years
* Currently taking Suboxone
* ASA (American Society of Anesthesiology) physical score 1-3
* Able to provide a signed informed consent
* General anesthesia (either endotracheal intubation or laryngeal mask airway) or MAC (monitored anesthesia care) without the use of regional anesthesia

Exclusion Criteria:

* Known allergic reactions to Dsuvia and its excipients
* Severe respiratory illness including exacerbation of asthma attack
* Significant intraoperative hemodynamic instability
* Use of Regional anesthesia techniques

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naum Shaparin, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson TA, Quaye ANA, Ward EN, Wilens TE, Hilliard PE, Brummett CM. To Stop or Not, That Is the Question: Acute Pain Management for the Patient on Chronic Buprenorphine. Anesthesiology. 2017 Jun;126(6):1180-1186. doi: 10.1097/ALN.0000000000001633. PMID 28511196
- [Background] Degenhardt L, Bucello C, Mathers B, Briegleb C, Ali H, Hickman M, McLaren J. Mortality among regular or dependent users of heroin and other opioids: a systematic review and meta-analysis of cohort studies. Addiction. 2011 Jan;106(1):32-51. doi: 10.1111/j.1360-0443.2010.03140.x. Epub 2010 Nov 4. PMID 21054613
- [Background] Johnson RE, Fudala PJ, Payne R. Buprenorphine: considerations for pain management. J Pain Symptom Manage. 2005 Mar;29(3):297-326. doi: 10.1016/j.jpainsymman.2004.07.005. PMID 15781180
- [Background] Alford DP, Compton P, Samet JH. Acute pain management for patients receiving maintenance methadone or buprenorphine therapy. Ann Intern Med. 2006 Jan 17;144(2):127-34. doi: 10.7326/0003-4819-144-2-200601170-00010. PMID 16418412
- [Background] Hansen HB, Siegel CE, Case BG, Bertollo DN, DiRocco D, Galanter M. Variation in use of buprenorphine and methadone treatment by racial, ethnic, and income characteristics of residential social areas in New York City. J Behav Health Serv Res. 2013 Jul;40(3):367-77. doi: 10.1007/s11414-013-9341-3. PMID 23702611
- [Background] Roberts DM, Meyer-Witting M. High-dose buprenorphine: perioperative precautions and management strategies. Anaesth Intensive Care. 2005 Feb;33(1):17-25. doi: 10.1177/0310057X0503300104. PMID 15957687
- [Background] Heel RC, Brogden RN, Speight TM, Avery GS. Buprenorphine: a review of its pharmacological properties and therapeutic efficacy. Drugs. 1979 Feb;17(2):81-110. doi: 10.2165/00003495-197917020-00001. PMID 378645
- [Background] Claxton AR, McGuire G, Chung F, Cruise C. Evaluation of morphine versus fentanyl for postoperative analgesia after ambulatory surgical procedures. Anesth Analg. 1997 Mar;84(3):509-14. doi: 10.1097/00000539-199703000-00008. PMID 9052292
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Felden L, Walter C, Harder S, Treede RD, Kayser H, Drover D, Geisslinger G, Lotsch J. Comparative clinical effects of hydromorphone and morphine: a meta-analysis. Br J Anaesth. 2011 Sep;107(3):319-28. doi: 10.1093/bja/aer232. Epub 2011 Aug 5. PMID 21841049
- [Background] Minkowitz HS, Leiman D, Melson T, Singla N, DiDonato KP, Palmer PP. Sufentanil Sublingual Tablet 30 mcg for the Management of Pain Following Abdominal Surgery: A Randomized, Placebo-Controlled, Phase-3 Study. Pain Pract. 2017 Sep;17(7):848-858. doi: 10.1111/papr.12531. Epub 2017 Feb 10. PMID 27781372
- [Background] Jove M, Griffin DW, Minkowitz HS, Ben-David B, Evashenk MA, Palmer PP. Sufentanil Sublingual Tablet System for the Management of Postoperative Pain after Knee or Hip Arthroplasty: A Randomized, Placebo-controlled Study. Anesthesiology. 2015 Aug;123(2):434-43. doi: 10.1097/ALN.0000000000000746. PMID 26079801
- [Background] Ringold FG, Minkowitz HS, Gan TJ, Aqua KA, Chiang YK, Evashenk MA, Palmer PP. Sufentanil sublingual tablet system for the management of postoperative pain following open abdominal surgery: a randomized, placebo-controlled study. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):22-30. doi: 10.1097/AAP.0000000000000152. PMID 25318408
- [Background] W.M. Tvetenstrand CD, Reduced Opioid Use and Reduced Time in the Postanesthesia Care Unit Following Preoperative Administration of Sublingual Sufentanil in an Ambulatory Surgery Setting., J Clin Anesth Pain Manag. 4 2.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled into the Control (Standard of Care) arm prior to study termination. As such, zero participants were identified in the corresponding categories for the Control (Standard of Care) arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalence
Description: Evaluate the total amount of morphine equivalence (MME) in the perioperative period (defined as combined total opioid used intra-op and in the PACU).
Time Frame: During day of surgery
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Fit to Discharge From the PACU (Post-Anesthesia Care Unit)
Description: How much time did subject take to become considered 'fit to discharge?'
Time Frame: During stay in PACU, up until discharge from PACU
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Need for Additional Opioids Following Surgery
Description: A measure of how any additional opioids subjects were administered
Time Frame: PACU stay to 24 hours post hospital discharge
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Take the First Additional Opioid
Description: Average time for administration of first additional opioid.
Time Frame: 24 hours post hospital discharge
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Adverse Events in the PACU
Description: Make note of nausea, vomiting, itching, hypotension, dizziness that occur while in PACU
Time Frame: During PACU stay, up until discharge from PACU
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Events Post Discharge From PACU
Description: Make note of nausea, vomiting, itching, hypotension, dizziness that occur within 24 hours after being discharged from PACU
Time Frame: 24 hours
Population: Data was not collected/aggregated. As such there was no data analysis for this terminated study.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Intraoperative period through 24 hours following discharge from PACU - an average of 24-48 hours.
Description: No participants were enrolled into the Control (Standard of Care) arm prior to study termination. As such, zero participants were identified as having been 'at risk' in the denominator for the Control (Standard of Care) arm.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT04716413/Prot_SAP_000.pdf